CLINICAL TRIAL: NCT03020472
Title: U19 Year 6: Kinetics of B-Cell Responses to Live, Attenuated Influenza Vaccine (LAIV) in Young Children Two Years of Age, SLVP016
Brief Title: Kinetics of B-Cell Responses to Live, Attenuated Influenza Vaccine (LAIV) in Young Children Two Years of Age
Acronym: SLVP016
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to low enrollment
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Philip Grant, Assistant Professor of Medicine (Infectious Diseases), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SU-15086; U19AI057229 (NIH)
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Influenza
Keywords: Live, attenuated influenza vaccine; Children
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2008-2009 FluMist LAIV (Intranasal) (Experimental): 2008-2009 FluMist LAIV (Intranasal) Seasonal live, attenuated influenza vaccine
  Interventions: Biological: 2008-2009 FluMist LAIV (Intranasal)

INTERVENTIONS:
Biological: 2008-2009 FluMist LAIV (Intranasal) — 2008-2009 FluMist vaccine delivered intranasally

SUMMARY:
This pilot study will investigate B-cell responses following vaccination with live, attenuated influenza vaccine (LAIV) in healthy children 2 years of age from blood samples taken at designated time points before and after vaccination.

DETAILED DESCRIPTION:
This is an exploratory study to determine the peripheral antibody secreting cell response during Days 5-13 after immunization with live, attenuated influenza vaccine (LAIV).

Investigators hoped to enroll 27 healthy children, 2 years of age who had not had any prior LAIV or trivalent inactivated vaccine (TIV) within the past 2 years. Due to low enrollment, the study was halted. Due to the limited number of samples, no analysis was performed.

ELIGIBILITY:
Inclusion Criteria

1. Otherwise healthy children, aged 24-35 months of age, inclusive.
2. Parent(s) or guardian(s) willing to sign informed consent.
3. Availability for follow-up for the planned duration of the study.
4. Acceptable medical history by screening evaluation and brief clinical assessment.
5. Able to understand and comply with planned study procedures

Exclusion Criteria

1. Prior vaccination with LAIV.
2. TIV vaccination during two prior influenza vaccine seasons
3. Known prior MD diagnosis of, or hospitalization for influenza
4. History of asthma, active/recurrent wheezing or reactive airways disease
5. History of immunodeficiency
6. Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease; diabetes mellitus; moderate to severe kidney impairment.
7. Known underlying medical conditions (e.g. hemoglobinopathy, congestive heart failure) predisposing to influenza complications.
8. Household contact with immunodeficiency due to disease, medication or radiation
9. Child receiving aspirin therapy or aspirin-containing therapy
10. History of Guillain-Barré syndrome
11. Malignancy, other than squamous cell or basal cell skin cancer
12. Autoimmune disease
13. Use of immunosuppressive medication. Corticosteroid nasal sprays are permissible.
14. Use of antiviral agents against Influenza A and/or B (such as Tamiflu, Relenza, Flumodine, Symmetrel) less than 48 hours before and/or less than two weeks after administration of FluMist.
15. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow-up or hospitalization during the preceding year.
16. Use of investigational agents within 30 days prior to study
17. Receipt of blood products or immunoglobulin in the past 6 months
18. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment
19. Acute febrile illness on the day of vaccination
20. Known allergies to any component of the vaccine, including eggs or egg products, gentamicin, gelatin,or arginine, or known life-threatening reactions to previous influenza vaccinations.
21. Concurrent participation in other investigational protocols or receipt of an investigational product within the previous 30 days or planned receipt of an investigational product within 28 days following the last immunization dose.
22. Any condition that, in the opinion of the investigator, might interfere with study objectives

Ages: 24 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry B Greenberg, MD, Principal Investigator — Stanford University; Xiaosong He, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 2008-2009 FluMist LAIV (Intranasal): Seasonal live, attenuated influenza vaccine (LAIV)
  2008-2009 FluMist LAIV (Intranasal): 2008-2009 FluMist vaccine delivered intranasally
Period: Overall Study
Arm/Group | 2008-2009 FluMist LAIV (Intranasal)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 2008-2009 FluMist LAIV (Intranasal)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.4 (0.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received Influenza Vaccine
Time Frame: Day 0 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | 2008-2009 FluMist LAIV (Intranasal)
Number analyzed (Participants) | 6
Participants | 6

2. Secondary Outcome: Number of Participants With Related Adverse Events
Time Frame: Day 0 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | 2008-2009 FluMist LAIV (Intranasal)
Number analyzed (Participants) | 6
Participants | 0

3. Other Pre Specified Outcome: Post- Immunization B- Cell Response
Description: Identify peak of the post-immunization B-cell responses following vaccination with live, attenuated influenza vaccine (LAIV)
Time Frame: 5-13 days post immunization
Population: Due to the low enrollment, the study was terminated and analysis was not performed.
Arm/Group | 2008-2009 FluMist LAIV (Intranasal)
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: PBMC Samples Will be Tested by Flow Cytometry to Determine the Percentage of Influenza-specific Antibody Cells That Are CD27+CD38+CD19+ Plasmablasts and by ELISPOT.
Time Frame: Day 0 to Day 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 2008-2009 FluMist LAIV (Intranasal)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No